CLINICAL TRIAL: NCT02605317
Title: Use of whatsApp Messenger (a Messaging Program for Smart Phones) in Communication Between Consulting Physicians and the Emergency Physicians: A Retrospective Observational Study
Brief Title: Use of WhatsApp for Communication Between Consulting Physicians and the Emergency Physicians
Acronym: whatsapp
Status: Completed | Type: Observational
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Principal Investigator, Adiyaman University Research Hospital
Other Study IDs: ADYU
Record Dates: First submitted 2015-11-11; First posted 2015-11-16 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Consultation
Keywords: Emergency Physicians; Consulting Physicians; WhatsApp

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: WhatsApp — Consultations used WhatsApp Messenger
  Other Names: A smart phone application

SUMMARY:
The aim of this study is to determinate outcomes of WhatsApp Messenger (a messaging program for smart phones) usage for Communication Between Consulting Physicians and the Emergency Physicians.

DETAILED DESCRIPTION:
Effective communication between consulting physicians and the emergency physicians is critical for patients in the emergency department. WhatsApp Messenger (a messaging program for smart phones), is the most commonly used for communication in at present. WhatsApp Messenger is the most globally popular messaging application. Also, it has been started to be used for communication in healthcare. The aim of this study is to determinate outcomes of WhatsApp Messenger usage for communication between consulting and the emergency physicians.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years

Exclusion Criteria:

* Patients who were not known the reason of admission to Emergency Service
* Patients who were not determined consulting Physicians' arrival duration to emergency department
* Patients who were not known the outcomes of consultation
* Patients transferred other hospitals from Emergency Service
* Patients who were not determined the time of consultation call

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were consulted with whatsApp and who were admitted to Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Examine outcomes of consultations generated with WhatsApp from data obtained by the recording data in the WhatsApp messenger program | six month
  Patients' demographic data (date of birth/age and gender), date of consultation, time of consultation calls, patients' reason of admission to Emergency Service, consulting Physicians' arrival duration to emergency department, outcomes of consultation, date of discharge from Emergency Service were noted by an assistant blinded to the study.

SECONDARY OUTCOMES:
Examine demographic data in consultations generated with WhatsApp from data obtained by the recording data in the WhatsApp messenger program | six month
  Patients' demographic data (date of birth/age and gender), date of consultation and patients' data such as imagine, voice, writing and laboratory results sent with WhatsApp were noted by an assistant blinded to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gulacti, Principal Investigator — Adiyaman University of Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)

REFERENCES:
- [Background] Astarcioglu MA, Sen T, Kilit C, Durmus HI, Gozubuyuk G, Kalcik M, Karakoyun S, Yesin M, Zencirkiran Agus H, Amasyali B. Time-to-reperfusion in STEMI undergoing interhospital transfer using smartphone and WhatsApp messenger. Am J Emerg Med. 2015 Oct;33(10):1382-4. doi: 10.1016/j.ajem.2015.07.029. Epub 2015 Jul 31. PMID 26299691
- [Background] Montag C, Blaszkiewicz K, Sariyska R, Lachmann B, Andone I, Trendafilov B, Eibes M, Markowetz A. Smartphone usage in the 21st century: who is active on WhatsApp? BMC Res Notes. 2015 Aug 4;8:331. doi: 10.1186/s13104-015-1280-z. PMID 26238512
- [Background] Veneroni L, Ferrari A, Acerra S, Massimino M, Clerici CA. [Considerations on the use of WhatsApp in physician-patient communication and relationship]. Recenti Prog Med. 2015 Jul;106(7):331-6. doi: 10.1701/1940.21090. Italian. PMID 26228724
- [Background] Drake TM, Claireaux HA, Khatri C, Chapman SJ. WhatsApp with patient data transmitted via instant messaging? Am J Surg. 2016 Jan;211(1):300-1. doi: 10.1016/j.amjsurg.2015.04.004. Epub 2015 May 28. No abstract available. PMID 26092444